CLINICAL TRIAL: NCT02641392
Title: A Phase 3, Long-term Active Treatment Extension Study of Mongersen (GED-0301) in Subjects With Crohn's Disease
Brief Title: A Long-term Active Treatment Study of Mongersen (GED-0301) in Subjects With Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by Sponsor following a recommendation from external DMC based on lack of emerging benefit; there were no new emergent safety findings
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GED-0301-CD-004
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; GED 0301; Mongersen; Safety; Irritable Bowel Disease
MeSH Terms: conditions — Crohn Disease; Irritable Bowel Syndrome | interventions — GED0301

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- GED-0301 (160 mg) followed by Placebo intermittent 160 mg (Experimental): GED-0301 160 mg once daily (QD) for 12 weeks, followed by alternating Placebo (PBO) QD for 4 weeks with GED 0301 160 mg QD for 4 weeks, up to 208 weeks, if the subject previously received Placebo in the prior GED-0301 Study
  Interventions: Drug: GED-0301
- Intermittent GED-0301 160 mg and placebo (Experimental): Alternating GED-0301 160 mg once daily (QD) for 4 weeks with placebo (PBO) QD for 4 weeks, up to 208 weeks, depending on previous response in the prior GED-0301 study
  Interventions: Drug: GED-0301; Other: Placebo
- Intermittent placebo and GED-0301 40 mg (Experimental): Alternating PBO once daily (QD) for 4 weeks with GED-0301 40 mg QD for 4 weeks with, up to 208 weeks, depending on previous response in the prior GED-0301 study
  Interventions: Drug: GED-0301; Other: Placebo
- Continuous GED-0301 40 mg (Experimental): GED-0301 40 mg once daily (QD) for up to 208 weeks
  Interventions: Drug: GED-0301
- Intermittent placebo and GED-0301 160 mg (Experimental): Alternating PBO QD for 4 weeks with GED-0301 160 mg QD for 4 weeks, through Week 208
  Interventions: Drug: GED-0301; Other: Placebo

INTERVENTIONS:
Drug: GED-0301 — Mongersen
  Other Names: Mongersen
Other: Placebo — Placebo
  Arms: Intermittent GED-0301 160 mg and placebo; Intermittent placebo and GED-0301 160 mg; Intermittent placebo and GED-0301 40 mg

SUMMARY:
The purpose of this study is to assess long-term safety data of GED-0301 for a period of up to 208 weeks in adult subjects (i.e., ≥ 18 years of age) who participated in the core Phase 3 GED-0301-CD-002 and GED-0301-CD-003 studies and adolescent subjects (i.e., 12 to 17 years of age) who participated in the core Phase 3 GED-0301-CD-003 study. Although all subjects will receive active treatment, this study is double-blinded for the entire 208 weeks for the purpose of preserving the blind of the subject's treatment allocation in the initial, core Phase 3 GED-0301 study.

The GED-0301-CD-003 trial was not initiated; see detailed description.

DETAILED DESCRIPTION:
This is a long-term active treatment study in patients with Crohn's disease (CD). Subjects who met the early escape criteria in Study GED-0301-CD-002, or subjects who completed Study GED-0301-002 or GED-0301-003, may be eligible for this study. Primary objective is to assess long-term safety of GED 0301. Additional efficacy and patient reported outcomes will be explored.

There are 5 possible treatment groups for GED-0301-CD-002 Subjects (Groups 1-5). There are 3 possible treatment groups for GED-0301-CD-003 subjects (Groups 1-3). Treatment is assigned based on clinical improvement achieved or not achieved from the core GED-0301 study.

1. continuous GED-0301 160 mg once daily for 12 weeks, followed by alternating placebo once daily for 4 weeks with GED-0301 160 mg once daily for 4 weeks, through Week 208;
2. alternating GED-0301 160 mg once daily for 4 weeks with placebo once daily for 4 weeks, through Week 208;
3. alternating placebo once daily for 4 weeks with GED-0301 160 mg once daily for 4 weeks, through Week 208;
4. continuous GED-0301 40 mg once daily through Week 208;
5. alternating placebo once daily for 4 weeks, followed by GED-0301 40 mg once daily for 4 weeks, through Week 208.

The GED-0301-CD-003 trial was not initiated; the GED-0301 program was terminated; no safety findings were noted.

ELIGIBILITY:
Inclusion Criteria for Adult Subjects:

Subjects must satisfy the following criteria to be screened and enrolled in the study:

* Male or female ≥ 18 years of age.
* Subject must have participated in the GED-0301-CD-002 or GED 0301 CD 003 study.
* Subject must use protocol approved contraception.

Inclusion Criteria for Adolescent Subjects:

Adolescent subjects must satisfy the following criteria to be screened and enrolled in the study

* Male or female 12 to 17 years of age.
* Subject must have participated in the GED 0301 CD 003 study.
* Subject is able to swallow the IP tablets.
* Subject must use protocol approved contraception.

Exclusion Criteria for Adult and Adolescent Subjects:

The presence of any of the following will exclude a subject from screening and enrollment:

* Subject had experienced a serious adverse event (SAE) related to the investigational product while participating in the previous Phase 3 GED-0301 study.
* Subject has initiated biologic agents, such as TNF-α blockers or integrin antagonists.
* Subject is pregnant or breastfeeding.
* Subject has developed a known hypersensitivity to oligonucleotides, GED 0301 or any ingredient in the investigational product.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Rossiter, MD, Study Director — Celgene
Locations (231):
- United States (23):
  - Medical Associates Research Group Inc., San Diego, California
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Health Science Research Center, LLC, Pratt, Kansas
  - Via Christi Research a division of Via Christi Hospitals Wichita Inc, Wichita, Kansas
  - Gastroenterology Associates LLC, Baton Rouge, Louisiana
  - Metropolitan Gastroenterology, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan PLC, Wyoming, Michigan
  - Ehrhardt Clinical Research LLC, Belton, Missouri
  - Columbia University Medical Center, New York, New York
  - Trial Management Associates LLC, Wilmington, North Carolina
  - ClinSearch LLC, Chattanooga, Tennessee
  - Texas Clinical Research Institute LLC, Arlington, Texas
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - Texas Digestive Disease Consultants - Southlake, Flower Mound, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Sagact Pllc, San Antonio, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - The Vancouver Clinic, Vancouver, Washington
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Centre For Digestive Diseases, Five Dock, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Monash Medical Centre Clayton, Bentleigh East
- Austria (7):
  - LKH Universitaetsklinikum Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - KH der Barmherzigen Bruder Linz, Linz
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - KH der Barmherzigen Brüder St.Veit an der Glan, Sankt Veit an der Glan
  - Krankenanstalt Rudolfstiftung Wien, Wein
  - AKH Medizinische Universitat Wien, Wein
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - UZ Leuven, Leuven
  - CHU Sart Tilman, Liège
- Bulgaria (7):
  - MHAT Kaspela EOOD, Plovdiv
  - MHAT Ruse AD, Rousse
  - Second MHAT Sofia AD, Sofia
  - City Clinic UMHAC EOOD, Sofia
  - UMHAT Sv Ivan Rilski EAD, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL EAD, Sofia
  - MHAT Doverie AD, Sofia
- Canada (16):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - South Edmonton Gastroenterology, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - GI Research Institute, Vancouver, British Columbia
  - PerCuro Clinical Research, Victoria, British Columbia
  - Brandon Medical Arts Clinic, Brandon, Manitoba
  - McMaster University Health Sciences Center, Hamilton, Ontario
  - London Health Science Center U. Hospital, London, Ontario
  - LHSC Victoria Hospital, London, Ontario
  - Montfort Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Digestive Disease Associates Inc, Vaughan, Ontario
  - Medicine Professional Corporation, Waterloo, Ontario
  - Centre de sante et de services sociaux Champlain Charles Le Moyne, Greenfield Park, Quebec
  - McGill University Health Centre Glen Site Royal Victoria Hospital, Montreal, Quebec
- Clinical Hospital Centre Osijek, Osijek, Croatia
- Czechia (4):
  - Fakultni nemocnice u sv Anny v Brne, Brno
  - Hepato-Gastroenterologie HK, Hradec Králové
  - PreventaMed, Olomouc
  - CCBR Prague CZ, Prague
- Denmark (6):
  - Aarhus Universitetshospital, Aahus C
  - Alborg Universitets Hospital, Aalborg
  - Nordsjaellands Hospital Frederikssund, Frederikssund
  - Herlev Hospital, Herlev
  - Koge Sygehus, Køge
  - Regionshospitalet Silkeborg, Silkeborg
- France (15):
  - CHU Amiens Hopital Sud, Amiens
  - CHU Besancon Hopital Jean Minjoz, Besançon
  - CHU Tours Hopital Trousseau, Chambray-lès-Tours
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - CHU Nantes Hotel Dieu, Nantes
  - CHU Nice Hopital de lArchet 2, Nice
  - Groupe Hospitalier Sud Hopital Haut Leveque USN, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Reims Hopital Robert Debre, Reims
  - CHU Rennes Hopital Pontchaillou, Rennes
  - CHU Saint Etienne Hopital Nord, Saint-Etienne
  - CHU Strasbourg Hopital Hautepierre, Strasbourg
  - CHU de Toulouse Hopital Rangueil, Toulouse
  - Hopital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (24):
  - Charite Universitaetsmedizin Berlin Campus Benjamin Franklin, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Krankenhaus Waldfriede e V, Berlin
  - Berufsgenossenschaftliches Universitaetsklinikum Bergmannsheil GmbH, Bochum
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Universitaetsklinikum Halle Saale, Halle
  - Asklepios Klinik Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Praxis fuer Gastroenterologie Dr Ehehal Dr Helmstaedter, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - University Leipzig, Leipzig
  - EUGASTRO GmbH, Leipzig
  - Medizinisches Zentrum Klinikum Lueneburg, Lüneburg
  - Klinikum Mannheim GmbH Universitaetsklinikum, Mannheim
  - Klinikum der Universitaet Muenchen, München
  - Gastro Campus Research, Münster
  - Staedtisches Klinikum Braunschweig gGmbH Standort Salzdahlumer, Niedersachsen
  - Universitaetsklinikum Regensburg, Regensburg
  - Universitaetsklinikum Ulm, Ulm
- Greece (4):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens Evangelismos, Athens
  - Athens Medical Center, Athens
  - University General Hospital of Patras, Rio Patras
- Hungary (8):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem AOK, Budapest
  - Endomedix Diagnosztikai Kozpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szent Pantaleon Korhaz Rendelointezet Dunaujvaros, Dunaújváros
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Clinfan Szolgaltato Kft, Szekszárd
- Israel (11):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center Department of Hematology, Tel Aviv
  - The Baruch Padeh MC, Poriya, Tiberias
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (12):
  - Azienda Ospedaliera Universitaria Policlinico Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Policlinico G Martino, Messina
  - Fondazione IRCCS CA Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Vincenzo Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Universita Campus Bio Medico di Roma, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Istituto Clinico Humanitas, Rozzano (MI)
  - IRCCS Policlinico San Donato, San Donato Milanese
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo FG
- Latvia (2):
  - Digestive Diseases Center Gastro, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Netherlands (6):
  - VU Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Radboudumc, Nijmegen
  - Zuyderland Medisch Centrum, Sittard-Geleen
  - St. Elisabeth Ziekenhuis, Tilburg
- Norway (2):
  - Akershus universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus Rikshospitalet, Oslo
- Poland (5):
  - Niepubliczny Zaklad Opieki Zdrowotnej POLIMEDICA, Kielce
  - Indywidualna Praktyka Lekarska Maciej Zymla, Knurów
  - SPZOZ Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej - Centralny Szpital Weteranow, Lodz
  - Centrum Medyczne Medyk, Rzeszów
  - Endoskopia Sp. z o.o., Sopot
- Portugal (2):
  - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira Guimaraes, Guimarães
- Romania (3):
  - S.C MedLife S.A, Bucharest
  - CMI Dr. Tirnaveanu Amelita, Oradea
  - Centrul de Gastroenterologie Dr. Goldis, Timișoara
- Russia (8):
  - TSBIH Territorial Clinical Hospital, Krasnoyarsk
  - SBHI of NN region RCH of NN n.a. N.A.Semashko, Nizhny Novgorod
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - FSBI Scientific Research Institute of Physyology and Basic Medicine under the SB of RAMS, Novosibirsk
  - Evromedservis, Pushkin
  - SEIHPE Rostov State Medical University of MoH of RF, Rostov-on-Don
  - SPb SBIH City Hospital # 26, Saint Petersburg
  - NonState Healthcare Institution Central Clinical Hospital, Samara station JSC Russian Railways, Samara
- Serbia (3):
  - Clinical Center Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta, Banská Bystrica
  - Alian s.r.o., Bardejov
  - Gastroeneterologicka ambulancia MUDr. Peter Hegyi s.r.o., Malacky
  - Fakultna nemocnica Nitra, Nitra
  - KM Management, spol. s r.o., Nitra
  - GASTRO I., s.r.o., Prešov
- South Korea (10):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Hanyang University Guri Hospital, Guri-si
  - CHA Bundang Medical Center CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Corporacion Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Miguel Servet, Zaragoza
- Danderyds Sjukhus AB, Stockholm, Sweden
- Crohn-Colitis Zentrum Bern Gemeinschaftspraxis Balsiger Seibold und Partner, Bern, Switzerland
- Turkey (Türkiye) (9):
  - Ankara University Medical Faculty, Ankara
  - Yeditepe University Medical School Hospital, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Istanbul
  - Acibadem Fulya Hospital, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Istanbul Medeniyet Uni Goztepe Training&Res Hosp, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli Derince Training and Research Hospital, Kocaeli
- Ukraine (9):
  - RCI Chernivtsi Regional Clinical Hospital Dept of Surgery Bukovinian SMU, Chernivtsi
  - CI of PH Kharkiv CCH #2, Kharkiv
  - Treatment-Diagnostic Center of Private Enterprise of PMF Atsynus, Kirovohrad
  - Ukrainian-German Antiulcer Gastroenterological Center BYK-Kyiv LLC, Kyiv
  - Kyiv City Clinical Hospital #1, Kyiv
  - SI Republican Clinical Hospital of the MOHU Dept of Gastroenterology O.O.Bogomolets NMU, Kyiv
  - CI Odesa Regional Clinical Hospital, Odesa
  - Ternopil City Communal Emergency Medical Care Hospital, Ternopil
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhya
- United Kingdom (10):
  - Royal Devon and Exeter Hospital Wonford, Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Hull Royal Infirmary, Hull
  - Royal London Hospital, London
  - St Marys Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Nottingham University Hospitals Queens Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford
  - Royal Shrewsbury Hospital, Shrewsbury

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 310 adult participants who had previously participated in the main study GED-0301-CD-002 were enrolled at 167 study sites in 29 countries.
Pre-assignment Details: Includes participants with Crohn's disease who had previously participated in the main study GED-0301-CD-002 through Week 12 at minimum and completed participation through the last treatment visit at Week 52, or met the "early escape criteria" and were discontinued beginning at Week 12 through Week 52.
Groups:
- GED-0301 40 mg 4 Weeks Alt: Participants received alternating placebo daily for 4 weeks and GED-0301 40 mg daily for 4 weeks, up to week 208
- GED-0301 40 mg: Participants received continuous GED-0301 40 mg daily, up to week 208.
- GED-0301 160 mg 4 Weeks Alt: Participants received one of three dose regimens up to week 208:
  1) alternating placebo daily for 4 weeks and GED-0301 160 mg daily for 4 weeks or (2) alternating GED-0301 160 mg daily for 4 weeks and placebo daily for 4 weeks or (3) GED-0301 160 mg daily for 12 weeks, followed by alternating placebo daily for 4 weeks and GED-0301 160 mg daily for 4 weeks
Period: Overall Study
Arm/Group | GED-0301 40 mg 4 Weeks Alt | GED-0301 40 mg | GED-0301 160 mg 4 Weeks Alt
Started | 4 | 13 | 293
Completed | 0 | 0 | 0
Not Completed | 4 | 13 | 293
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 17
Not completed — Adverse Event | 0 | 1 | 25
Not completed — Study Terminated by Sponsor | 4 | 12 | 144
Not completed — Lack of Efficacy | 0 | 0 | 101
Not completed — Miscellaneous | 0 | 0 | 3
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Long Term Active Population
Groups:
- Total: Total of all reporting groups
Arm/Group | GED-0301 40 mg 4 Weeks Alt | GED-0301 40 mg | GED-0301 160 mg 4 Weeks Alt | Total
Number analyzed (Participants) | 4 | 13 | 293 | 310
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (12.34) | 41.8 (14.21) | 38.1 (12.30) | 38.2 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 136 | 145
  Male | 1 | 7 | 157 | 165
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 0 | 3 | 10 | 13
  Black or African American | 0 | 0 | 3 | 3
  White | 4 | 9 | 264 | 277
  Not Collected or Reported | 0 | 1 | 10 | 11
  Other | 0 | 0 | 4 | 4
Duration of Crohn's Disease [Mean (Standard Deviation); unit: Years] | 7.25 (6.529) | 9.25 (6.307) | 10.56 (8.503) | 10.46 (8.396)
Baseline Crohn's Disease Activity (CDAI) Score [Mean (Standard Deviation); unit: units on a scale] — The Crohn's Disease Activity Index (CDAI) is used to quantify the signs and symptoms of Crohn's disease and the effect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450.
  units on a scale | 316.9 (96.90) | 309.2 (43.10) | 307.5 (62.74) | 307.7 (62.33)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events From Week 0 to Week 208
Description: A TEAE was defined as any adverse event (AE) occurring or worsening on or after the first treatment of GED-0301 and up to 28 days after the last GED- 0301 dose or the last follow-up date, whichever occurred earlier. A serious AE = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs was assessed by the investigator and based on the following scale; Mild = asymptomatic or mild symptoms; clinical or diagnostic observations only; Moderate = Symptoms cause moderate discomfort; Severe (could be non-serious or serious) = symptoms causing severe discomfort/pain.
Time Frame: From the first day of GED-0301 until 28 days after the last dose of IP; maximum treatment duration was 16.1 weeks in the GED-0301 40 mg Alt dose; 16.3 weeks in the GED 40 mg continuous dose and 56.1 weeks in the GED-0301 160 mg Alt dose
Population: Safety population includes participants who were received at least one dose of GED-0301. Participants were included in the group corresponding to the treatment regimen they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- GED 40 mg 4 Weeks Alt: Participants received alternating placebo daily for 4 weeks and GED-0301 40 mg daily for 4 weeks, up to week 208
Arm/Group | GED 40 mg 4 Weeks Alt | GED-0301 40 mg | GED-0301 160 mg 4 Weeks Alt
Number analyzed (Participants) | 4 | 13 | 293
Participants
  Any TEAE | 1 | 6 | 189
  Any Drug-Related TEAE | 0 | 1 | 43
  Any Severe TEAE | 0 | 0 | 38
  Any Serious TEAE (SAE) | 1 | 0 | 41
  Any Serious Drug-Related TEAE | 0 | 0 | 4
  Any TEAE Leading to IP Interruption | 0 | 0 | 7
  Any TEAE Leading to IP Withdrawal | 0 | 1 | 27
  Any TEAE Leading to Death | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the first day of GED-0301 up tol 28 days after the last dose of GED-0301.
Description: Maximum treatment duration was 16.1 weeks in the GED-0301 40 mg Alt dose; 16.3 weeks in the GED 40 mg continuous dose and 56.1 weeks in the GED-0301 160 mg Alt dose
Arm/Group | GED-0301 40 mg 4 Weeks Alt | GED-0301 40 mg | GED-0301 160 mg 4 Weeks Alt
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/13 | 1/293
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/13 | 41/293
Other Adverse Events (participants affected / at risk) | 1/4 | 6/13 | 92/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GED-0301 40 mg 4 Weeks Alt (N=4) | GED-0301 40 mg (N=13) | GED-0301 160 mg 4 Weeks Alt (N=293)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 2
ANAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 2
ANAL STENOSIS (Gastrointestinal disorders) | 0 | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 0 | 12
ILEAL STENOSIS (Gastrointestinal disorders) | 0 | 0 | 5
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 | 0 | 1
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 | 0 | 4
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
SUBILEUS (Gastrointestinal disorders) | 0 | 0 | 2
DROWNING (General disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 1
HYPERTHERMIA (General disorders) | 0 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 0 | 1
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 3
APPENDICITIS (Infections and infestations) | 0 | 0 | 1
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1
GROIN ABSCESS (Infections and infestations) | 0 | 0 | 1
INFECTIOUS COLITIS (Infections and infestations) | 0 | 0 | 1
PERIRECTAL ABSCESS (Infections and infestations) | 0 | 0 | 2
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 | 0 | 1
PULMONARY SEPSIS (Infections and infestations) | 0 | 0 | 1
SALMONELLOSIS (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
VULVAL ABSCESS (Infections and infestations) | 0 | 0 | 1
ANASTOMOTIC ULCER HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 1
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 1 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 1
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
VESICAL FISTULA (Renal and urinary disorders) | 0 | 0 | 1
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GED-0301 40 mg 4 Weeks Alt (N=4) | GED-0301 40 mg (N=13) | GED-0301 160 mg 4 Weeks Alt (N=293)
CARDIAC VALVE DISEASE (Cardiac disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 29
ANAL FISTULA (Gastrointestinal disorders) | 0 | 1 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 0 | 1 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1 | 30
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 0
ILEAL STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 20
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 1 | 0 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2 | 27
HEADACHE (Nervous system disorders) | 0 | 0 | 16

LIMITATIONS AND CAVEATS:
Following a recommendation by the Data Monitoring Committee (DMC), the study was terminated early by Celgene on 19 Oct 2017 due to a lack of emerging benefit; no emergent safety findings were noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
.Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT02641392/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT02641392/SAP_001.pdf